CLINICAL TRIAL: NCT00068588
Title: A Phase 2 Study of GTI-2040 (NSC 722929) in Combination With Capecitabine in Metastatic Breast Cancer
Brief Title: GTI-2040 and Capecitabine in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02827; PHII-46; N01CM62209 (NIH); CDR0000327757 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2013-01

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — GTI2040; Capecitabine

ARMS (1):
- Treatment (GTI-2040, capecitabine) (Experimental): Patients receive GTI-2040 IV continuously on days 1-15 of the first course and days 1-14 of all subsequent courses. Patients also receive oral capecitabine twice daily on days 2-15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: GTI-2040; Drug: capecitabine

INTERVENTIONS:
Biological: GTI-2040 — Given IV
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda

SUMMARY:
This phase II trial is studying how well giving GTI-2040 together with capecitabine works in treating patients with metastatic breast cancer. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. GTI-2040 may help capecitabine kill more tumor cells by making them more sensitive to the drug

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate and response duration to combination therapy with GTI-2040 and capecitabine in the treatment of metastatic breast cancer.

II. To safely evaluate the toxicity of this drug combination and schedule in this patient population by first using a lower dose followed by escalation.

III. To determine pharmacokinetic data on plasma levels of GTI-2040 in this patient population.

IV. To investigate potential molecular markers of ribonucleotide reductase inhibition and fluoropyrimidine metabolism in this patient population treated with the combination of GTI-2040 and capecitabine.

OUTLINE: This is a multicenter study.

Patients receive GTI-2040 IV continuously on days 1-15 of the first course and days 1-14 of all subsequent courses. Patients also receive oral capecitabine twice daily on days 2-15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic adenocarcinoma of the breast
* Patients must have measurable disease, defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients must have progressed on at least one but no more than two prior chemotherapy regimens for metastatic disease; patients must not have received prior capecitabine or 5-fluorouracil; patients with hormone-sensitive tumors should have received hormone treatment and any prior number of hormonal agents will be allowed; patients with tumors that overexpress HER-2/neu (3+ by immunohistochemistry or amplified by fluorescent in situ hybridization) should have received herceptin, either in the adjuvant or metastatic setting, unless there is a contraindication to herceptin therapy; all prior therapies must have been completed 4 weeks before treatment
* Life expectancy of greater than 3 months
* ECOG performance status =< 2 (Karnofsky >= 50%)
* Leukocytes >= 3,000/μL
* Absolute neutrophil count >= 1,500/μL
* Platelets >= 100,000/μL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min
* Patients must have completed radiation treatment > 4 weeks prior to study entry; previously radiated area(s) must not be the only site of disease
* All major surgical procedures must be completed > 4 weeks prior to study entry; placement of vascular access device or tissue biopsy will not be considered major surgery
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients must agree to the placement of a central venous catheter in order to receive the continuous infusion treatment

Exclusion Criteria:

* Patients with only non-measurable disease, defined as all other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions, which include the following:

  * bone lesions
  * leptomeningeal disease
  * ascites
  * pleural/pericardial effusion
  * inflammatory breast disease
  * lymphangitis cutis/pulmonis
  * abdominal masses that are not confirmed and followed by imaging techniques
  * cystic lesions
* Patients who have had chemotherapy, hormone therapy, or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents; patients may not have received prior GTI-2040
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GTI-2040 or to capecitabine or 5-fluorouracil
* Patients requiring anticoagulant therapy; low-dose anticoagulant (warfarin 1 mg per day) for the primary prophylaxis of venous catheter-associated thrombosis is permitted
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because GTI-2040 and capecitabine have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with GTI-2040 and capecitabine, breastfeeding should be discontinued if the mother is treated
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with GTI-2040 or other agents administered during the study; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Chew, Principal Investigator — City of Hope Medical Center
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1st 3 pts treated on arm 2. If 0/3 DLTs, escalate to arm 3. If 1/3 DLTs on arm 2, 3 more pts on arm 2. If 1/6 DLTs on arm 2, escalate to arm 3.If at most 1/6 DLTs on arm 3, MTD declared. If more than 1/6 DLTs on arm 3, then de-escalated to arm 2. If at most 1/6 DLTs on arm 2, MTD declared. If more than 1/6 DLTs on arm 2, then de-escalate to arm 1.
Groups:
- Arm 1: Capecitabine 800 mg/m2 BID for 14 days on days 2-15 of each 21 day cycle +GTI-2040 civ infusion 185 mg/m2/day on days 1-15 of cycle 1 and days 1-14 of each subsequent cycle,
- Arm 2: Capecitabine 1000 mg/m2 BID for 14 days on days 2-15 of each 21 day cycle +GTI-2040 civ infusion 185 mg/m2/day on days 1-15 of cycle 1 and days 1-14 of each subsequent cycle,
- Arm 3: Capecitabine 1250 mg/m2 BID for 14 days on days 2-15 of each 21 day cycle +GTI-2040 civ infusion 185 mg/m2/day on days 1-15 of cycle 1 and days 1-14 of each subsequent cycle,
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 0 | 3 | 21
Completed | 0 | 3 | 17
Not Completed | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Poor KPS | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 0 | 3 | 21 | 24
Age, Continuous [Median (Full Range); unit: years] |  | 63 [42 to 64] | 52 [39 to 74] | 53 [39 to 74]
Gender [Number; unit: participants]
  Female |  | 3 | 21 | 24
  Male |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 21 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose Determined by Dose-limiting Toxicities
Description: 1st 3 pts will be treated on arm 2. If 0/3 DLTs observed, the dose will be escalated to arm 3. If 1/3 DLTs onserved on arm 2, 3 more pts will be treated on arm 2. If no additional DLTs are observed on arm 2, the dose will be escalated to arm 3. If at most 1/6 DLTs observed on arm 3, arm 3 will be considered the MTD. If more than 1/6 DLTs observed on arm 3, the dose will be de-escalated to arm 2. If at most 1/6 DLTs observed on arm 2, arm 2 will be considered the MTD. If more than 1/6 pts on arm 2 experience a DLT, the dose will be de-escalated to arm 1. The remaining pts will be treated on arm 1 as the MTD, unless more than 1/6 DLTs, in which case the study will stop. DLT is defined as any grade III or IV non-hematologic toxicity (incl. diarrhea w\ adequate antidiarrheal treatment & hydration & nausea/vomiting w\ maximal antiemetic prophylaxis, as per protocol) or grade IV hematologic toxicity. DLT will be based on the 1st course of treatment according to the revised NCI CTC v 2.0
Time Frame: 21 days
Measure: Number; unit: Patients experiencing DLT
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 3 | 6
Patients experiencing DLT |  | 0 | 0

2. Primary Outcome: Response Rate of a Combination of GTI-2040 and Capecitabine
Description: Following the dose escalation step, additional patients will be accrued at the MTD and evaluated for disease response using RECIST v1.0 criteria. Patients with confirmed complete or partial response are considered to have responded favorably to treatment.The sample size and early stopping for futility was governed by a two stage Optimum design suggested by Simon. It was assumed that a true response rate less than 25% would not warrant further study of this agent. It was also assumed that a response rate of 45% would be considered promising. In the first stage (following the dose escalation step), 15 evaluable patients were treated. Four or fewer observed responses, would stop accrual, while 5 or more observed would continue accrual for an additional 12 patients during the second stage of the study. Ten or more responses out of 27 patients will be considered evidence warranting further study of the regimen providing toxicity and survival also appear favorable.
Time Frame: Up to 6 years
Population: Response Rate was only assessed at the determined MTD. Additional patients were accrued to determine treatment efficacy at the MTD.
Measure: Number; unit: percentage of patients responding
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 15
percentage of patients responding |  |  | 20

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 5.5 year period in which patients were actively treated.
Description: There was one death six days after treatment stopped possibly related to treatment described as "somnolence/depressed level of consciousness". "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 2/3 | 6/21
Other Adverse Events (participants affected / at risk) | 3/3 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 2 (N=3) | Arm 3 (N=21)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Infection NOS (Infections and infestations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 2 (N=3) | Arm 3 (N=21)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (5) | 19 (64)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Conjunctival disorder (Eye disorders) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 5 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3)
Incontinence NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 4 (6)
Nausea (Gastrointestinal disorders) | 2 (4) | 5 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 0 (0) | 3 (4)
Fatigue (General disorders) | 3 (7) | 16 (54)
Fever (General disorders) | 0 (0) | 3 (3)
General symptom (General disorders) | 1 (1) | 11 (11)
Injection site reaction (General disorders) | 1 (2) | 0 (0)
Oedema NOS (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 5 (8)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4) | 14 (49)
Alkaline phosphatase increased (Investigations) | 1 (2) | 12 (37)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 17 (82)
Creatinine increased (Investigations) | 1 (1) | 1 (2)
Hypercholesterolemia (Investigations) | 0 (0) | 1 (3)
INR increased (Investigations) | 0 (0) | 2 (3)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (2)
Leukopenia (Investigations) | 2 (5) | 16 (72)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Lymphopenia (Investigations) | 0 (0) | 11 (29)
Neutrophil count decreased (Investigations) | 2 (3) | 15 (57)
(Investigations) | 1 (2) | 2 (6)
Platelet count decreased (Investigations) | 0 (0) | 12 (48)
Weight gain (Investigations) | 0 (0) | 1 (2)
Weight loss (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 12 (31)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 11 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 13 (48)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 7 (14)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 9 (35)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (4)
Taste alteration (Nervous system disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (3)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (9)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (55)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (5)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
In the first stage of the two stage Optimum design, following the dose escalation step, 3 of 15 patients responded for a response rate of 20%. A response rate of less than 25% would not warrant further study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less